CLINICAL TRIAL: NCT04703348
Title: Pilot Study on the Assessment of Motor Imaging Skills in Patients With Complex Regional Pain Syndrome (CRPS)
Brief Title: The Complex Regional Pain Syndrome (CRPS) is a Chronic Pain Condition. This is a Preliminary Study to Explore and Test Clinical Hypothesis. They Suppose That CRPS Patients Have Impairment in Their Mental or Motor Imagery Abilities.
Acronym: ImagNimes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: LOCAL/2020/MO-01; 2020-A02281-38 (Other: ANSM)
Record Dates: First submitted 2021-01-07; First posted 2021-01-11 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2022-11

CONDITIONS: Complex Regional Pain Syndromes; Musculoskeletal Pain Disorder; Healthy
Keywords: complex regional pain syndromes; motor imagery; mental imagery; MIQ-RS; Pilot study; comparison groups; CRPS
MeSH Terms: conditions — Complex Regional Pain Syndromes; Collagen Diseases

STUDY DESIGN:
Intervention Model Description: 3 groups with different healthcare conditions are compared in motor imagery capacities
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Healthy patients (Other): Healthy patients take the MIQ-RS during about 40 minutes : about 20 minutes for the assessment of the right side and about 20 minutes for the left side
  Interventions: Diagnostic Test: Motor imagery Questionnaire - Revised Second (MIQ-RS)
- Complex regional pain syndrome patients (Other): Complex regional pain syndrome patients take the MIQ-RS during about 40 minutes : about 20 minutes for the assessment of the right side and about 20 minutes for the left side
  Interventions: Diagnostic Test: Motor imagery Questionnaire - Revised Second (MIQ-RS)
- Musculoskelettal disorders patients (Other): Musculoskelettal disorders patients take the MIQ-RS during about 40 minutes : about 20 minutes for the assessment of the right side and about 20 minutes for the left side
  Interventions: Diagnostic Test: Motor imagery Questionnaire - Revised Second (MIQ-RS)

INTERVENTIONS:
Diagnostic Test: Motor imagery Questionnaire - Revised Second (MIQ-RS) — Patients fulfill a questionnaire measuring individuals capacities to realize mental imagery. For more facilities and less risk of bias, the MIQ-RS was written on an online version with questions recorded in audio format. No official cut-off exists but studies seem to prove that people with :
  * a score less than 48/98 are unable to do motor imagery
  * a score between 49 and 73/98 have disturbed motor imagery capacities
  * a score more than 74/98 have normal motor imagery capacities.

SUMMARY:
Medical functional imagery seems to demonstrate that patients suffering from complex regional pain syndrome (CRPS) have cortical modifications that alter their motor (or mental) imagery capacities. Nowadays, the use of motor imagery exercises are used in conventional rehabilitation treatments. But, in clinical practice, no study has verified if patients with CRPS desmonstrate problems in their motor imagery capacities. The MIQ-RS (Motor Imagery Questionnaire - Revised Second) is a valid, reliable and translated into French questionnaire to measure patients' capacities to do mental imagery. In this study, we compare 3 groups of 50 patients : healthy patients, patients with CRPS and patients with musculoskeletal disorder without CRPS. Every patient will take the MIQ-RS for the right and left body side. We hypothesis that patients with CRPS have more deficit than the 2 others to realise motor imagery.

ELIGIBILITY:
Inclusion Criteria:

* Patient with French healthcare affiliation
* Adult patient (> 18 years old)
* Patient with bachelor degree minimum
* Patient practicing less than 150 minutes of moderate to intense physical activity per week

Specific Inclusion Criteria for CRPS group :

* Patient followed in the Evaluation and Treatment pain center (University Hospital of Nimes)
* Patient with secondary CRPS due to a traumatism or a surgery

Specific Inclusion Criteria for Musculoskeletal group :

* Patient with musculoskelettal disorder on a limb (upper or lower)
* Patient followed in the University Hospital of Nimes

Non inclusion Criteria :

* Patient who participates in another category 1 research
* Patient in a exclusion period in another study
* Patient under legal protection, under guardianship or under curatorship
* Patient for whom it is impossible to give clear information.
* Pregnant, parturient or breastfeeding patient.
* Patient with amputation on one of his limb
* Patient with visual cecity
* Patient who has already practiced mental imagery
* Patient with neurological impairment
* Patient with chronic low back pain and fibromyalgia

Specific non inclusion criteria for Musculoskeletal group and healthy group :

-Patient with CRPS

Specific non inclusion Criteria for CRPS group :

* Secondary CRPS to CVA (cerebrovascular accident)
* Patient receiving lymph node block treatment between the inclusion visit and the follow-up visit

Specific non inclusion Criteria for Musculoskeletal Disorder group :

* Patient with secondary musculoskeletal disorder to a CVA

Exclusion criteria :

* Questionnaire MIQ-RS not completed or non respect with the research protocol
* pathology discovered incompatible with the study criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 129 (Actual)
Dates: Start 2021-01-12 (Actual); Primary Completion 2022-10-30 (Actual); Study Completion 2022-10-30 (Actual)

PRIMARY OUTCOMES:
Motor imagery capacities on the affected side for CRPS group and musculoskelettal disorder group. | Day 1
  Taking the MIQ-RS for 1 side, during about 20 minutes The questionnaire includes 14 questions : 7 for kinesthesic motor imagery and 7 for visual motor imagery For less bias, the questionnaire was recorded in audio for each of the 14 questions on an online assessment.
  No official cut-off exists but studies seem to prove that people with :
  * a score less than 48/98 are unable to do motor imagery
  * a score between 49 and 73/98 have disturbed motor imagery capacities
  * a score more than 74/98 have normal motor imagery capacities.

SECONDARY OUTCOMES:
Motor imagery capacities between affected side and unaffected side | Day 1
  Taking the MIQ-RS for 1 side, during about 20 minutes The questionnaire includes 14 questions : 7 for kinesthesic motor imagery and 7 for visual motor imagery For less bias, the questionnaire was recorded in audio for each of the 14 questions on an online assessment.
  No official cut-off exists but studies seem to prove that people with :
  * a score less than 48/98 are unable to do motor imagery
  * a score between 49 and 73/98 have disturbed motor imagery capacities
  * a score more than 74/98 have normal motor imagery capacities.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Nimes, Nîmes, Gard, France

REFERENCES:
- [Result] Cohen-Aknine G, Mottet D, Homs AF, Mura T, Jedryka F, Dupeyron AF. Explicit Motor Imaging Abilities Are Similar in Complex Regional Pain Syndrome, Chronic Limb Pain and Healthy Individuals: A Cross-Sectional Study. J Pain Res. 2025 Apr 11;18:1949-1961. doi: 10.2147/JPR.S494546. eCollection 2025. PMID 40236719
- See also: Related Info — https://rsds.org/wp-content/uploads/2015/05/ICC-Pollard.pdf
- See also: Related Info — https://link.springer.com/article/10.1007/s11724-014-0368-x